CLINICAL TRIAL: NCT02756052
Title: Enhancing Laparoscopic Skill Acquisition and Retention With Transcranial Direct-current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Patrick Ciechanski, PhD Candidate (Neurosciences), University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REB15-2443
Record Dates: First submitted 2016-03-30; First posted 2016-04-29 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Laparoscopic Surgical Procedures
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Medical Student - Sham tDCS (Sham Comparator): Participants: 1st to 3rd year medical students from the Cumming School of Medicine (University of Calgary).
  Device: Sham tDCS. 45 second ramp up to 1milliamp, 60 second current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Sham Transcranial direct-current stimulation
- General Surgery Resident - Sham tDCS (Sham Comparator): Participants: 1st to 5th year general surgery residents from the Cumming School of Medicine (University of Calgary).
  Device: Sham tDCS. 45 second ramp up to 1milliamp, 60 second current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Sham Transcranial direct-current stimulation
- Medical Student - Anodal tDCS (Experimental): Participants: 1st to 3rd year medical students from the Cumming School of Medicine (University of Calgary).
  Device: Anodal tDCS. 45 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Anodal Transcranial direct-current stimulation
- General Surgery Resident - Anodal tDCS (Experimental): Participants: 1st to 5th year general surgery residents from the Cumming School of Medicine (University of Calgary).
  Device: Anodal tDCS. 45 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Interventions: Device: Anodal Transcranial direct-current stimulation

INTERVENTIONS:
Device: Anodal Transcranial direct-current stimulation — NeuroConn Direct-Current Stimulator. Anodal tDCS: 45 second ramp up to 1milliamp, 20 minute current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Other Names: Anodal tDCS
  Arms: General Surgery Resident - Anodal tDCS; Medical Student - Anodal tDCS
Device: Sham Transcranial direct-current stimulation — NeuroConn Direct-Current Stimulator. Sham tDCS: 45 second ramp up to 1milliamp, 60 second current hold at 1milliamp, 45 second ramp down to 0milliamp. Anode positioned 2cm posterior to the left primary motor cortex, and the cathode over the contralateral supraorbital area.
  Other Names: Sham tDCS
  Arms: General Surgery Resident - Sham tDCS; Medical Student - Sham tDCS

SUMMARY:
Recent changes in medical training environments and restrictive work-hour regulations have greatly impacted trainees, limiting the number of opportunities to gain proficiency in procedural skills. Reports suggest that medical residents lack confidence in their ability to perform certain medical procedures, and program directors often do not believe their residents can operate independently in major procedures. Simulator based task training (SBTT) has provided a safe and ethically appropriate method of skill acquisition but training opportunities remain limited. Methods to enhance motor learning during these training opportunities have not been described. Transcranial direct-current stimulation (tDCS) is an emerging form of non-invasive brain stimulation that has been shown to improve motor learning. tDCS has been shown to enhance increasingly complex skill acquisition. The investigators propose to examine if tDCS can improve the acquisition and retention of laparoscopic surgical skill. The investigators propose a double blind, sham-controlled randomized trial applying tDCS during evidence-based SBTT of medical students and surgical residents, to determine if brain stimulation can enhance training effects and long-term skill acquisition. Even a modest enhancement carries the potential to transform medicosurgical skills training.

DETAILED DESCRIPTION:
Rationale: Recent changes in medical training environments have resulted in many trainees lacking sufficient opportunity to acquire specific skills necessary for their specialty. New methods to enhance the acquisition and retention of medical and surgical skills are required to ensure the quality of the future physician workforce. Transcranial direct-current stimulation (tDCS) is an emerging method of non-invasive brain stimulation that has been show to safely enhance motor learning in adults and children. Even a modest enhancement of acquisition and retention of medical-surgical skill with tDCS carries the potential to accelerate skill training for health care providers, thereby contributing to greater training efficiency and improved patient outcomes.

Objectives: The objective of this study is to assess whether tDCS can enhance the acquisition and retention of laparoscopic surgical ability.

Ethics:This study has been approval by the University of Calgary Research Ethics Board

Design: Randomized, double blind, sham-controlled trial to evaluate the ability of tDCS to enhance learning and retention of laparoscopic skills.

Transcranial Direct-Current Stimulation: The tDCS methods used are based on best-available evidence and practices, and will be applied in a standardized fashion by experienced investigators. Anodal tDCS will be delivered through saline-soaked sponge electrodes using a NeuroConn Direct-Current Stimulator (NeuroConn, Ilmenau, Germany). The anode will be centered 2cm posterior to the left primary motor cortex (localized using the 10-20 EEG System), with the cathode over the contralateral supraorbital area. Both anodal and sham tDCS groups will have the current ramped up to 1milliamp over 30 seconds. In the anodal tDCS group, the current will be held for 20 minutes. In the sham tDCS condition, the current will be held for only 60 seconds (no changes in cortical excitability) followed by a 30 second ramp-down.

Participants: Medical students (years 1-3) and general surgery residents (Post-Graduate Year 1-5) from the Cumming School of Medicine (University of Calgary) will be recruited. To ensure comparable baseline skills, trainees will be excluded if they have undergone formal laparoscopic training in the past 3 months (medical students only).

Sample size calculations are based on the performance measures for the pattern cutting score, determined through pilot studies (discussed below). Based on a two-fold greater improvement in score at post-training, power of 90% and type-1 error of 0.05, the investigators estimate a sample size of a minimum of 48 participants (n=24 per stimulation condition, with an equal number of residents and medical students per arm).

Study Design: A short questionnaire will be completed to determine demographic characteristics, including: gender, age, level of training, date of last completed Fundamentals of Laparoscopic Surgery course (if applicable), how many times participants have performed laparoscopic surgery on a patient, how many times participants have performed laparoscopic tasks on a laparoscopic simulator, how often participants play video games, and how often participants play a musical instrument.

Participants will be recruited at the Advanced Technical Skills and Simulation Laboratory (University of Calgary) and be oriented to the workspace. Participants will complete laparoscopic task training on a laparoscopic box trainer (Fundamentals of Laparoscopic Surgery Trainer System, Limbs & Things Inc, Georgia, USA) consisting of an optic camera, laparoscopic instruments, and a monitor that displays the field of view. The optic camera view will be recorded for retroactive scoring. Participants will view a standardized laparoscopic training video, created by an expert in laparoscopic surgery, demonstrating two Fundamentals of Laparoscopic Surgery (FLS) tasks that will be performed using the simulator: a peg-transfer (A) and pattern cutting task (B). The peg-transfer task requires the use of two dissectors to transfer six rings to pegs on the opposite end of the pegboard, and back to the original location. The pattern-cutting task involves a 10x10cm piece of gauze with a 4cm-diameter circle pre-drawn in the middle that is placed at the center of the work-board. Participants are required to use a dissector and endoscopic scissors to cut the marked circle, freeing it from the surrounding unmarked gauze. A time score will be calculated by subtracting the completion time in seconds from the task cut-off time of 300 seconds. An error score will be calculated for each tasks as either: the percentage of pegs that could not be transferred due to being dropped outside of the field of view (i.e. 1 of 6 pegs lost = 17 second penalty), or the percentage area deviation of cutting a perfect circle. A total score is calculated by subtracting the error score from the time score. These two FLS tasks represent skills that require bimanual (peg-transfer) or unimanual (pattern cutting) abilities. Furthermore, these two tasks were chosen as scores correlate with training level, and are predictive of intraoperative performance.

Participants will complete task A followed by task B, establishing baseline skill. Tasks will be recorded and scored retroactively, blinded to group allocation, to quantify time and error scores. Participants will be computer randomized to receive sham or active tDCS. Participants will perform the two FLS tasks in an interleaved manner (ABAB), a paradigm suggested to enhance laparoscopic skill acquisition, with eight training repetitions of each task. Following the final training block, the tDCS electrodes will be removed, and a final task evaluation will be performed for both task A and B. The Purdue Pegboard Test (PPT) will be performed at baseline and post-training to examine unilateral hand function, serving as a safety measure. Six weeks following the training the participants will return to assess retention of laparoscopic skill, with a single repetition of task A and B. Emerging evidence suggests that a significant decay in laparoscopic skill is present six weeks following training. The amount of laparoscopic practice between the training day and follow-up will be factored for residents, to ensure that standard training remains uninterrupted.

Data Analysis: Mean change in each outcome from baseline to post-training to follow-up will be compared between tDCS and sham (two-way repeated-measure ANOVA for factors "stimulation type" and "evaluation time point"). Two-way repeated-measures ANOVA for factors "stimulation type" and "training block" will explore the interaction between tDCS and training with or without feedback for each outcome. Any decay in PPT score in either sham or anodal tDCS groups will be evaluated using a paired-tDCS. Medical students and specialty residents will be evaluated independently. Level of training of residents will be factored retroactively into our analysis.

ELIGIBILITY:
Inclusion Criteria:

* Medical student or general surgery residents
* Informed consent

Exclusion Criteria:

* Diagnosis of a developmental, neurological or neuropsychiatric disorder
* Taking neuropsychotropic medication
* Has an irremovable implanted metal object in the head
* Has a pacemaker or other implanted electrical device
* Pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Fundamentals of Laparoscopic Surgery pattern cutting task total score | Baseline and Immediately Post-Training
  A "baseline trial" will be performed, followed by 8 consecutive "training trials", immediately followed by a "post-training trial".
  A total score is calculated by subtracting the error score from the time score. A time score will be calculated by subtracting the completion time in seconds from the task cut-off time of 300 seconds. An error score will be calculated as the percentage area deviation of cutting a perfect circle.
Change in Fundamentals of Laparoscopic Surgery peg transfer task total score | Baseline and Immediately Post-Training
  A "baseline trial" will be performed, followed by 8 consecutive "training trials", immediately followed by a "post-training trial".
  A total score is calculated by subtracting the error score from the time score. A time score will be calculated by subtracting the completion time in seconds from the task cut-off time of 300 seconds. An error score will be calculated as the percentage of pegs that could not be transferred due to being dropped outside of the field of view (i.e. 1 of 6 pegs lost = 17 second penalty).

SECONDARY OUTCOMES:
Retention of Fundamentals of Laparoscopic Surgery pattern cutting task total score | 6 Weeks following Training
  Retention of skill will be examined 6 weeks following the training session. The score will be calculated as outlined in the primary outcome measure.
Retention of Fundamentals of Laparoscopic Surgery peg transfer task total score | 6 Weeks following Training
  Retention of skill will be examined 6 weeks following the training session. The score will be calculated as outlined in the primary outcome measure.

OTHER OUTCOMES:
Change in Purdue Pegboard Test score | Baseline and Immediately Post-Training
  The Purdue Pegboard Test will be performed at baseline and immediately post-training, as a safety measure of general hand function. Participants will have 30 seconds to place as many pegs as they using the left or right hand. The test will be repeated 3 times with each hand. The "Change in Purdue Pegboard Test score" will be calculated by taking an average of the score of 3 repetitions per hand.
Visual Analog Scale for tDCS-sensations | Baseline and Immediately Post-Training
  The sensations of "itching, burning, tingling, discomfort, and pain" will be ranked by the participant using a numeric visual analog scale. Participants rank each sensation independently on a scale from 0-10, where "0" refers to "sensation not present", "5" refers to "sensation was moderately tolerable" and "10" refers to "sensation was untolerable".

CONTACTS AND LOCATIONS:
Locations (1):
- Cumming School of Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis FR, Klingensmith ME. Issues in general surgery residency training--2012. Ann Surg. 2012 Oct;256(4):553-9. doi: 10.1097/SLA.0b013e31826bf98c. No abstract available. PMID 22964740
- [Background] Coleman JJ, Esposito TJ, Rozycki GS, Feliciano DV. Early subspecialization and perceived competence in surgical training: are residents ready? J Am Coll Surg. 2013 Apr;216(4):764-71; discussion 771-3. doi: 10.1016/j.jamcollsurg.2012.12.045. PMID 23521960
- [Background] Mattar SG, Alseidi AA, Jones DB, Jeyarajah DR, Swanstrom LL, Aye RW, Wexner SD, Martinez JM, Ross SB, Awad MM, Franklin ME, Arregui ME, Schirmer BD, Minter RM. General surgery residency inadequately prepares trainees for fellowship: results of a survey of fellowship program directors. Ann Surg. 2013 Sep;258(3):440-9. doi: 10.1097/SLA.0b013e3182a191ca. PMID 24022436
- [Background] Derossis AM, Fried GM, Abrahamowicz M, Sigman HH, Barkun JS, Meakins JL. Development of a model for training and evaluation of laparoscopic skills. Am J Surg. 1998 Jun;175(6):482-7. doi: 10.1016/s0002-9610(98)00080-4. PMID 9645777
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Reis J, Fritsch B. Modulation of motor performance and motor learning by transcranial direct current stimulation. Curr Opin Neurol. 2011 Dec;24(6):590-6. doi: 10.1097/WCO.0b013e32834c3db0. PMID 21968548
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Derived] Ciechanski P, Cheng A, Damji O, Lopushinsky S, Hecker K, Jadavji Z, Kirton A. Effects of transcranial direct-current stimulation on laparoscopic surgical skill acquisition. BJS Open. 2018 Mar 13;2(2):70-78. doi: 10.1002/bjs5.43. eCollection 2018 Apr. PMID 29951631